CLINICAL TRIAL: NCT02198053
Title: Effect of 180 mgTicagrelor Compared With 90 mg Ticagrelor on Platelet Reactivity in Patients Undergoing Elective PCI.
Brief Title: the Effect Between Platelet Reactivation and Antiplatelet Drugs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, quan li, associate chief physician, Beijing Anzhen Hospital
Other Study IDs: azliquan
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Drug Effect Disorder; Platelet Procoagulant Activity Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Platelet reactivity
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ticagrelor2: Ticagrelor with a loading dose of 180mg followed by 90 mg twice per day
- Ticagrelor1: Ticagrelor with a dose of 90mg followed by 90 mg twice per day .

SUMMARY:
Different antiplatelet drugs played various role in coronary artery disease. The mechanisms were unclear. Platelet reactivation maybe was one of major causes. Compared with clopidogrel, Ticagrelor is more powerful antiplatelet drug. However, because of increased bleeding and dyspnea risk, both loading double dose and following second dose time had potential risk and inconvenient in routine clinical work, especially in elective PCI of comparable stable patients in Chinese. The benefit and risk should be balanced in such patients. The investigators supposed loading single dose and followed by second routine time dose was superior to clopidogrel and safer than ticagrelor previously prescribed.

DETAILED DESCRIPTION:
All admission patients were divided into two groups, the first group were prescribed loading dose (180 mg) ticagrelor, the second group were prescribed with 90 mg ticagrelor. We measured both platelet activity and platelet reactivity using the LTA at baseline, pre-operation and post-operation. All bleeding or dyspnea events were recorded in hospital period.

Primary endpoints: platelet activity, platelet reactivity using the LTA and safety events were recorded in hospital period.

ELIGIBILITY:
Inclusion Criteria:

coronary artery disease, percutaneous coronary intervention

Exclusion Criteria:

high risk bleeding patient, allergic to the drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | 1 year
  LTA and TEG used to measure the effect of Platelet reactivity

CONTACTS AND LOCATIONS:
Overall Officials: LI QUAN, doctor, Study Director — Beijing Anzhen Hospital
Locations (1):
- Anzhen Hospital, Beijing, China